CLINICAL TRIAL: NCT03585647
Title: Effect of Anesthetics Used for Regional vs General vs Integrated Anesthesia on the Modulation of 'Stress-responsive' Genes Involved in the Metabolism and Cellular Detoxification
Brief Title: Anesthetic Methods and Gene Expression Profile
Acronym: GeSTA
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, RAlleva, PhD, University of Bologna
Other Study IDs: 12630
Record Dates: First submitted 2018-06-14; First posted 2018-07-13 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hip Arthroplasty
Keywords: General anesthesia; Regional anesthesia; Integrated anesthesia; Hip arthroplasty; Toxicological gene expression
MeSH Terms: interventions — Arthroplasty, Replacement, Hip; Hip Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be obtained from all enrolled patients. The samples will be collected in heparin tubes and peripheral blood mononuclear cell (PBMC) fraction will be isolated for total RNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GA-group: Patients undergoing elective hip arthroplasty included in the GA-group received general anesthesia. GA was induced by intravenous fentanyl (1 mcg/kg) and propofol (2 mg/kg), followed by vecuronium bromide (0.1 mg/kg) to facilitate tracheal intubation, then GA was maintained using a 50% air/oxygen mixture and sevoflurane.The end-tidal concentration of sevoflurane was adjusted to maintain heart rate and blood pressure values within 20% of baseline. Mechanical ventilation was regulated to maintain the end-tidal carbon dioxide partial pressure ranging between 4.3 and 5.1 kilopascal.
  Interventions: Procedure: hip arthroplasty
- RA-group: Patients undergoing elective hip arthroplasty included in the RA-group received regional anesthesia. Regional anaesthesia included continuous lumbar plexus block, performed by or under supervision of an experienced operator using a nerve stimulator (Stimulax, B. Braun) and Continued Peripheral Nerve Block Set.
  A total dose of 20 ml of 0.5% Levobupivacaine was administered at the time of catheter placement. Dural puncture was performed at the L3-L4 interspace using a 25-Gauge whitaker spinal needle (Becton-Dickinson, New Jersey, USA) with the midline approach using 3 ml of 0.5% Levobupivacaine.
  Interventions: Procedure: hip arthroplasty
- IA-group: Patients undergoing elective hip arthroplasty included in the IA-group received integrated anesthesia. The patients received regional anaesthesia (lumbar plexus block + spinal anaesthesia) as described protocol. General anaesthesia was induced by propofol 1% and a laryngeal mask airway of appropriate size was inserted. General anaesthesia and mechanical ventilation were maintained as standard protocol.
  Interventions: Procedure: hip arthroplasty

INTERVENTIONS:
Procedure: hip arthroplasty — Hip replacement is a surgery for people with severe hip damage. The most common cause of damage is osteoarthritis.
  Other Names: Hip prosthesis

SUMMARY:
The study will analyze differentially regulated genes involved in oxidative stress and toxicology in peripheral blood mononuclear cells (PBMCs) of patients who underwent arthroplasty under three different anesthetic methods. The investigator hypothesized that anesthesia procedures trigger toxicity, thus inducing changes in the messenger ribonucleic acid (mRNA) profile. The results may provide a more profound understanding of the molecular mechanism of anesthesia and in overcoming the adverse effects arising from their use.

DETAILED DESCRIPTION:
By using a computer-generated randomization table, hospitalized patients undergoing elective hip arthroplasty will be randomly consecutively allocated to receive general (GA group), regional (RA group), or integrated (IA group) anesthesia. Patients with contraindication to spinal anesthesia or lumbar catheter placement, as well as obese patients, with arterial hypertension not controlled by oral medication, severe pulmonary, cardiovascular, renal, hepatic, cerebrovascular, or psychiatric diseases will be excluded from the study.

Whole blood samples (10 mL) will be obtained from all enrolled patients at three time points: early morning on the operation day (T0), after surgery (T1) and third day (T2) after surgery. The samples will be collected in heparin tubes and PBMCs will be isolated and used for gene expression analysis. Serum obtained after blood centrifugation will be used for hematological and biochemical analysis such as glutamate oxaloacetate transaminase (GOT), glutamate-pyruvate transaminase (GPT), bilirubin (BIL), creatinine (CREA), creatine phosphokinase (CPK), hemoglobin (HB).

The sample size was determined according to Lee- Whitmore * and G*Power Ftest for ANOVA Fixed effects, omnibus, one-way (Lee ML, Whitmore GA. Stat Med. 2002;21: 3543-3570). Assuming a Poisson distribution for the expected value of the false-positive gene expression of the 9 chosen genes and fixing at 1 the maximum expected value for false positives E(R0) and considering all the 84 genes as not differentially expressed (G0=G=9), the probability α for any single gene among the G genes that are not differentially expressed is given by α=E(R_0 )/G=1/9=0.011, with the Bonferroni correction it becomes α_c=(0.011)/3=0.037. This is the type I error of a false positive expression. Moreover, considering as primary endpoint the fold increase of the gene expression, assuming a log-normal distribution with standard deviation of 0.7 which is typical of moderate-high gene expression and therefore a conservative one for the sample size determination and imposing a minimum difference on logarithmic scale among the 3 groups of 0.5 with a power of at least 0.8 and a Bonferroni corrected type I error α=0.05/3=0.0167 (which is smaller and then conservative, than the previous α_c) the minimum sample size(G*POWER)^ for each group is 30 patients, by considering a 10% of drop-out , the chosen sample size was 33 patients per group which leads to a total sample size of 99 patients.

^F tests - ANOVA: Fixed effects, omnibus, one-way Analysis: A priori: Compute required sample size Input: Effect size f = 0.7 α err prob = 0.0167 Power (1-β err prob) = 0.8 Number of groups = 3 Output: Noncentrality parameter λ = 14.7000000 Critical F = 4.7803455 Numerator df = 2 Denominator df = 27 Total sample size = 30 Actual power = 0.8009945

The normal distribution of continuous variables will be evaluated by Kolmogorov-Smirnov test. The Chi-square test will be used to evaluate categorical variables. The differences between groups will be evaluated by means of parametric ANOVA tests followed by Tukey test. Multiple regression analysis will be performed to evaluate the influence of biochemical parameters on gene expression in response to anesthetics considering confounding factors such as age, gender, BMI, smoking. Values of p <0.05 will be considered statistically significant. All tests will be performed using software (SPSS, Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologists Classification (ASA Class) = I-II.

Exclusion Criteria:

* American Society of Anesthesiologists Classification (ASA Class) > III
* contraindication to spinal anaesthesia or lumbar catheter placement
* arterial hypertension not controlled by oral medication
* severe pulmonary
* cardiovascular disease
* renal disease
* hepatic disease
* cerebrovascular disease
* psychiatric diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective hip arthroplasty
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2015-06-20 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Changes of Gene expression profile from baseline at time points | Gene expression will be evaluated in PBMCs at baseline (T0), up-30 min after surgery (T1) and on the third day (T2) after surgery.
  Effect of anesthesia techniques on the expression of genes indicative of stress and toxicity

SECONDARY OUTCOMES:
Relationship between deregulated genes and hepatic/renal cytotoxicity from baseline at time points | Biochemical analysis have been evaluated in blood collected at baseline (T0), up-30 min after surgery (T1) and on the third day (T2) after surgery.
  Multiple regression analysis of deregulated gene expression values (relative expression) and HB (mg/ml), hepatic markers such as GOT, GPT, BIL (mg/dl), and renal markers including CREA and CPK (mg/dl) will been performed. The results will be reported as coefficient of regression (r) with statistical significance p<0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Battista Borghi, MD, Study Director — Rizzoli Orthopaedic Institute
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual patient data (IPD) available

REFERENCES:
- [Result] Alleva R, Tomasetti M, Solenghi MD, Stagni F, Gamberini F, Bassi A, Fornasari PM, Fanelli G, Borghi B. Lymphocyte DNA damage precedes DNA repair or cell death after orthopaedic surgery under general anaesthesia. Mutagenesis. 2003 Sep;18(5):423-8. doi: 10.1093/mutage/geg013. PMID 12960410
- [Result] Borghi B, Casati A, Iuorio S, Celleno D, Michael M, Serafini PL, Alleva R. Effect of different anesthesia techniques on red blood cell endogenous recovery in hip arthroplasty. J Clin Anesth. 2005 Mar;17(2):96-101. doi: 10.1016/j.jclinane.2004.05.005. PMID 15809124
- [Result] Nakazato K, Yoshida Y, Takemori K, Kobayashi K, Sakamoto A. Expressions of genes encoding drug-metabolizing enzymes are altered after sevoflurane, isoflurane, propofol or dexmedetomidine anesthesia. Biomed Res. 2009 Feb;30(1):17-24. doi: 10.2220/biomedres.30.17. PMID 19265259
- [Result] Ishikawa M, Tanaka S, Arai M, Genda Y, Sakamoto A. Differences in microRNA changes of healthy rat liver between sevoflurane and propofol anesthesia. Anesthesiology. 2012 Dec;117(6):1245-52. doi: 10.1097/ALN.0b013e3182746676. PMID 23090150
- [Derived] Alleva R, Tognu A, Tomasetti M, Benassi MS, Pazzaglia L, van Oven H, Vigano E, De Simone N, Pacini I, Giannone S, Gagic S, Borghi R, Picone S, Borghi B. Effect of different anaesthetic techniques on gene expression profiles in patients who underwent hip arthroplasty. PLoS One. 2019 Jul 25;14(7):e0219113. doi: 10.1371/journal.pone.0219113. eCollection 2019. PMID 31344051